CLINICAL TRIAL: NCT01509677
Title: A 16-week, Randomized, Placebo-controlled, Double Blind, and Parallel Group Trial to Assess the Anti-inflammatory Effects of Roflumilast in Chronic Obstructive Pulmonary Disease
Brief Title: Trial to Assess the Anti-inflammatory Effects of Roflumilast in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO-2455-402-RD; 2011-000582-13 (EudraCT Number); U1111-1155-8767 (Registry Identifier: WHO); D7120C00003 (Other: Sponsor Identifier)
Record Dates: First submitted 2011-12-21; First posted 2012-01-13 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: Roflumilast; Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roflumilast (Active Comparator): 500 μg tablet, once daily, oral administration in the morning after breakfast
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): tablet, once daily, oral administration in the morning after breakfast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — 500 μg tablet, once daily, oral administration in the morning after breakfast
  Other Names: Daxas
  Arms: Roflumilast
Drug: Placebo — tablet, once daily, oral administration in the morning after breakfast
  Other Names: Placebo to Roflumilast
  Arms: Placebo

SUMMARY:
The objective of the Biopsy trial is to investigate the effect of roflumilast 500 µg tablets once daily versus placebo on inflammation parameters in bronchial biopsy tissue specimen and additional in sputum and blood serum. Also data on safety status will be obtained.

Patients to be included required to have moderate to severe COPD associated with chronic bronchitis. The total duration of this randomized, multicentre, phase III trial is 24 weeks maximum.

DETAILED DESCRIPTION:
This was a multicenter, double-blind, randomized, parallel group, phase 3 study. Patients included had a history of COPD (GOLD stage II-III, in Germany stage II only) with chronic productive cough.

There were 2 parallel treatment arms (placebo and roflumilast 500 μg once daily). A 1 to 1 randomization scheme was used, that is, patients were allocated to roflumilast 500 μg or placebo in equal proportions. Randomization was stratified by concomitant LABA use.

The total duration of this study was 24 weeks maximum per patient. The study consisted of the following periods:

* Single-blind placebo run-in period (6 weeks) with visits at Week -6 (visit 0 [V0]), Week -2 (V1), and Week 0 (V2, randomization visit), during which all patients received placebo.
* Double-blind treatment period (16 weeks) during which patients received either roflumilast or matching placebo with visits at Week 6 (V4), Week 14 (V5), and Week 16 (V6).

An additional visit (V3) within 2 weeks after bronchoscopy/bronchial biopsy was performed purely as a safety visit. The exact timing of this safety visit was to be determined by the investigator. Safety follow-up. All AEs were followed up to 30 days after the double-blind treatment period. An additional safety visit, V7, was scheduled within 2 weeks after the second bronchoscopy. The exact timing of the safety visit was to be determined by the investigator.

Patients were required not to take any food or drink overnight for at least 8 hours prior to returning to the study center for each visit. Patients were also asked to avoid strenuous exercise for 8 hours prior to each study visit and to avoid smoking for 4 hours prior to each study visit.

For visits where patients did not undergo blood collections or biopsies, the fasting requirement was only mandated if clinically indicated, per investigator judgment.

ELIGIBILITY:
Major Inclusion Criteria:

* Giving written informed consent
* History of COPD (according to GOLD 2009) for at least 12 months prior to baseline visit V0 associated with chronic productive cough for at least three months in each of the two years prior to baseline visit V0 (with other causes of productive cough excluded)
* Outpatients 40-80 years of age
* Post-bronchodilator 30% ≤FEV1 ≤80% predicted
* Post-bronchodilator FEV1/FVC ratio ≤70%
* Current or former smokers with smoking history ≥20 pack years

Main Exclusion Criteria:

• Criteria affecting the read-out parameters of the trial:

* Clinical instability, defined as experiencing a COPD exacerbation six months prior to V0
* An upper/lower respiratory tract infection which has not resolved four weeks prior to V0
* Diagnosis of asthma and/or other relevant lung disease
* Known alpha-1-antitrypsin deficiency
* Suspicion or diagnosis of a bleeding disorders irrespective of its pathophysiological mechanism
* Other protocol-defined exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (18):
- København NV, Denmark
- Germany (7):
  - Freiburg im Breisgau
  - Großhansdorf
  - Hanover
  - Heidelberg
  - Immenhausen
  - Kiel
  - Mainz
- Poland (3):
  - Bialystok
  - Krakow
  - Lodz
- Lund, Sweden
- United Kingdom (6):
  - Cottingham
  - Dafen
  - Leicester
  - London
  - Manchester
  - Norwich

REFERENCES:
- [Derived] Rabe KF, Watz H, Baraldo S, Pedersen F, Biondini D, Bagul N, Hanauer G, Gohring UM, Purkayastha D, Roman J, Alagappan VKT, Saetta M. Anti-inflammatory effects of roflumilast in chronic obstructive pulmonary disease (ROBERT): a 16-week, randomised, placebo-controlled trial. Lancet Respir Med. 2018 Nov;6(11):827-836. doi: 10.1016/S2213-2600(18)30331-X. Epub 2018 Sep 14. PMID 30224319
- See also: RO-2455-402-RD Updated Protocol v 6.0 (Amendment 12) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4560&filename=RO-2455-402-RD_ROBERT_Updated_Protocol_v6.0_(Amendment_12)_-_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- R500: Roflumilast 500 µg
- Placebo: Placebo to Roflumilast
Period: Overall Study
Arm/Group | R500 | Placebo
Started | 79 | 79
Completed | 76 | 73
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R500 | Placebo | Total
Number analyzed (Participants) | 79 | 79 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (8.23) | 62.5 (8.43) | 63.2 (8.34)
Age, Customized [Number; unit: Participants]
  Between 18 and 65 years | 37 | 46 | 83
  >=65 years | 42 | 33 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 60 | 61 | 121
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 77 | 77 | 154
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: Participants]
  Europe | 79 | 79 | 158

OUTCOME MEASURES:

1. Primary Outcome: Number of CD8+ Inflammatory Cells in Bronchial Biopsy Tissue.
Time Frame: 16 weeks
Population: The CD8+ cells count results in submucosa for the primary outcome were available for 117 patients at V2 (41 missing) and 114 patients at V6 (44 missing). The reason for missing samples was that the sample amount did not reach the minimal area requested per study protocol. See section 11.4.1 in CSR
Measure: Mean (Standard Deviation); unit: CD8+ cells count
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 49 | 46
CD8+ cells count | 442.4 (312.74) [0.82 to 1.30] | 427.1 (261.42)

2. Primary Outcome: Change in Number of CD8+ Inflammatory Cells in Bronchial Biopsy Tissue
Time Frame: Baseline to 16 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 49 | 46
cells/mm^2 | 13.4 (302.69) | 29.4 (298.88)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided test at 5% significant level; Test type: Superiority or Other; p = 0.7922, Poisson regression model — This is p-value testing significance of "treatment" effect
Statistical Analysis 2: Comparison: R500 vs Placebo; Test type: Superiority; p = 0.7917, Poisson regression model; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.82 to 1.30], Standard Error of Mean 0.120

3. Secondary Outcome: CD68+ Count in Biopsied Material (Submucosa)
Time Frame: 16 weeks
Population: The reason for missing samples was that the sample amount did not reach the minimal area requested per study protocol. See 11.4.7 in CSR
Measure: Mean (Standard Deviation); unit: CD68+ Count
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 49 | 46
CD68+ Count | 149.1 (113.91) | 124.4 (93.15)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided, 5% test; Test type: Superiority or Other; p = 0.7145, Poisson regression model — This is p-value testing significance of "treatment" effect

4. Secondary Outcome: CD68+ Cell Count in Biopsied Material (Submucosa): Poisson Regression (Ratio)
Description: CD68+ Cell Count in Biopsied Material (submucosa): Poisson regression (ratio). Clarification: Measure type described as "Number" refers to "Risk of each treatment group". It is not possible to select "risk" from this template so "number" was selected instead. This issue applies to similar variables reporting poisson regression.
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Number; unit: CD68+ Cell Count
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 49 | 46
CD68+ Cell Count | 126.8 (NA) | 121.6 (NA)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.7136, Poisson regression model; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.83 to 1.30], Standard Error of Mean 0.119

5. Secondary Outcome: Change From V2 to V6 in CD68+ Cell Count (Cells/mm^2) in Biopsied Material (Submucosa) (ITT)
Time Frame: Baseline and 16 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: CD68+ Cell Count (cells/mm^2)
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 49 | 46
CD68+ Cell Count (cells/mm^2) | 6.1 (10.99) | -5.3 (11.05)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.4606, ANCOVA; Mean Difference (Final Values) = 11.4, 95% CI [-19.2 to 42.1], Standard Error of Mean 15.45

6. Secondary Outcome: CD4+ Cell Counts in Biopsied Material (Submucosa):Poisson Regression Model
Description: CD4+ Cell Counts in biopsied Material (submucosa):poisson regression model. Clarification: Measure type "Number" refers to "Risk of each treatment group".
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Number; unit: CD4+ Cell Counts
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 48 | 46
CD4+ Cell Counts | 304.6 (NA) | 255.0 (NA)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.2744, Poisson regression model; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.87 to 1.64], Standard Error of Mean 0.194

7. Secondary Outcome: CD45+ Cell Counts in Biopsied Material (Submucosa):Poisson Regression Model
Description: CD45+ Cell Counts in biopsied Material (submucosa):poisson regression model. Clarification: Measure type "Number" refers to "treatment risk"
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Number; unit: CD45+ Cell Counts
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 49 | 46
CD45+ Cell Counts | 818.4 (NA) | 960.3 (NA)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.1128, Poisson regression model; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.70 to 1.04], Standard Error of Mean 0.086

8. Secondary Outcome: Neutrophils Cell Counts in Biopsied Material (Submucosa):Poisson Regression Model
Description: Neutrophils Cell Counts in biopsied Material (submucosa):poisson regression model. Clarification: Measure type "Number" refers to "Treatment risk"
Time Frame: Baseline to 14 weeks
Population: as for outcome 3
Measure: Number; unit: Neutrophils Cell Counts
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 49 | 46
Neutrophils Cell Counts | 118.6 (NA) | 127.7 (NA)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.6740, Regression, Linear; Poisson regression model; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.66 to 1.31], Standard Error of Mean 0.164

9. Secondary Outcome: CD8+ Cell Count in Biopsied Material (Bronchial Epithelium): Poisson Regression Model
Description: CD8+ Cell Count in biopsied material (Bronchial Epithelium): poisson regression model. Clarification: Measure Type "Number" refers to "Treatment risk"
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Number; unit: CD8+ Cell Count
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 41 | 37
CD8+ Cell Count | 422.1 (NA) | 505.3 (NA)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.0677, Poisson regression model; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.69 to 1.01], Standard Error of Mean 0.082

10. Secondary Outcome: CD68+ Cell Count in Biopsied Material (Bronchial Epithelium):Poisson Regression Model
Description: CD68+ Cell Count in biopsied material (Bronchial Epithelium):poisson regression model. Clarification: Measure type "Number" refers to "Treatment Risk"
Time Frame: 16 weeks
Population: as for outcome 3
Measure: Number; unit: CD68+ Cell Count
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 39 | 32
CD68+ Cell Count | 76.3 (NA) | 93.1 (NA)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.3566, Poisson regression model; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.54 to 1.25], Standard Error of Mean 0.177

11. Secondary Outcome: Change From V1 to V5 in Absolute Cell Count in Induced Sputum (10^6 Neutrophils/mL): Between-Treatment Difference
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 neutrophils/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 43 | 44
10^6 neutrophils/mL | 1.7181 (1.64471) | 0.0827 (1.61220)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2 sided 5% test; Test type: Superiority or Other; p = 0.4794, ANCOVA; Mean Difference (Final Values) = 1.6354, 95% CI 2-sided [-2.9429 to 6.2137], Standard Error of Mean 2.30185

12. Secondary Outcome: Change From V1 to V5 in Absolute Cell Count inInduced Sputum (10^6 Macrophages/mL): Between-Treatment Difference
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 macrophages/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 43 | 44
10^6 macrophages/mL | 0.1017 (0.23396) | -0.3710 (0.22970)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2 sided 5% test; Test type: Superiority or Other; p = 0.1541, ANCOVA; Mean Difference (Final Values) = 0.4727, 95% CI 2-sided [-0.1810 to 1.1264], Standard Error of Mean 0.32866

13. Secondary Outcome: Change From V1 to V5 in Absolute Cell Count inInduced Sputum (10^6 Eosinophils/mL): Between-Treatment Difference
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 eosinophils/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 43 | 44
10^6 eosinophils/mL | -0.0986 (0.02639) | -0.0360 (0.02585)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2 sided 5% test; Test type: Superiority or Other; p = 0.0927, ANCOVA; Mean Difference (Final Values) = -0.0626, 95% CI 2-sided [-0.1358 to 0.0106], Standard Error of Mean 0.03681

14. Secondary Outcome: Change From V1 to V5 in Absolute Cell Count inInduced Sputum (10^6 Lymphocytes/mL): Between-Treatment Difference
Time Frame: BAseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 lymphocytes/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 43 | 44
10^6 lymphocytes/mL | -0.0167 (0.01167) | -0.0060 (0.01141)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2 sided 5% test; Test type: Superiority or Other; p = 0.5175, ANCOVA; Mean Difference (Final Values) = -0.0107, 95% CI 2-sided [-0.0435 to 0.0220], Standard Error of Mean 0.01647

15. Secondary Outcome: Change From V1 to V5 in Differential Cell Count in Induced Sputum(10^6 Neutrophils/mL)
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 neutrophils/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 45 | 44
10^6 neutrophils/mL | 2.527 (2.3571) | 0.382 (2.3535)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5 % test; Test type: Superiority or Other; p = 0.5205, ANCOVA; Mean Difference (Final Values) = 2.146, 95% CI 2-sided [-4.466 to 8.757], Standard Error of Mean 3.3253

16. Secondary Outcome: Change From V1 to V5 in Differential Cell Count in Induced Sputum(10^6 Macrophages/mL)
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 macrophages/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 45 | 44
10^6 macrophages/mL | 0.315 (2.1328) | -0.826 (2.1316)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5 % test; Test type: Superiority or Other; p = 0.7052, ANCOVA; Mean Difference (Final Values) = 1.141, 95% CI 2-sided [-4.835 to 7.117], Standard Error of Mean 3.0057

17. Secondary Outcome: Change From V1 to V5 in Differential Cell Count in Induced Sputum(10^6 Eosinophils/mL)
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 eosinophils/m
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 45 | 44
10^6 eosinophils/m | -1.826 (0.5214) | -0.041 (0.5200)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5 % test; Test type: Superiority or Other; p = 0.0127, ANCOVA; Mean Difference (Final Values) = -1.867, 95% CI 2-sided [-3.324 to -0.409], Standard Error of Mean 0.7331

18. Secondary Outcome: Change From V1 to V5 in Differential Cell Count in Induced Sputum(10^6 Lymphocytes)/mL)
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: 10^6 lymphocytes)/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 45 | 44
10^6 lymphocytes)/mL | -0.137 (0.1332) | -0.086 (1.329)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5 % test; Test type: Superiority or Other; p = 0.7862, ANCOVA; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.423 to 0.321], Standard Error of Mean 0.1871

19. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Induced Sputum: Primary Parameters of Interest (FAS) (Alfa- 2-Macroglobulin (µg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: µg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 54 | 57
µg/mL | -0.32 (0.730) | -0.48 (0.700)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.8769, ANCOVA; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-1.84 to 2.15], Standard Error of Mean 1.005

20. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Induced Sputum: Primary Parameters of Interest (FAS) (IL-8 (pg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 54 | 56
pg/mL | -827.3 (1995.79) | -1538.4 (1941.08)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.7978, ANCOVA; Mean Difference (Final Values) = 711.1, 95% CI 2-sided [-4778.3 to 6200.5], Standard Error of Mean 2768.79

21. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Induced Sputum: Primary Parameters of Interest (FAS) (MMP Type 9 (ng/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 55 | 57
ng/mL | 80.1 (57.07) | -8.4 (55.44)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.2669, ANCOVA; Mean Difference (Final Values) = 88.5, 95% CI 2-sided [-68.6 to 245.6], Standard Error of Mean 79.26

22. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Induced Sputum: Primary Parameters of Interest (FAS) (MCP-1 (pg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 53 | 57
pg/mL | -95.2 (49.23) | -69.3 (46.93)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.7033, ANCOVA; Mean Difference (Final Values) = -25.9, 95% CI 2-sided [-160.3 to 108.5], Standard Error of Mean 67.78

23. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Induced Sputum: Primary Parameters of Interest (FAS) (TIMP-1 (ng/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 54 | 57
ng/mL | 25.87 (13.085) | -1.92 (12.551)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.1264, ANCOVA; Mean Difference (Final Values) = 27.79, 95% CI 2-sided [-7.97 to 63.55], Standard Error of Mean 18.039

24. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Induced Sputum: Primary Parameters of Interest (FAS) (VEGF (pg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 55 | 57
pg/mL | 253.1 (89.46) | -43.7 (86.84)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.0185, ANCOVA; Mean Difference (Final Values) = 296.8, 95% CI 2-sided [50.9 to 542.7], Standard Error of Mean 124.07

25. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Blood Serum: Primary Parameters of Interest (FAS) (Alfa-2-Macroglobulin (µg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: µg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 68 | 66
µg/mL | -0.05 (0.061) | -0.05 (0.062)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.9989, ANCOVA; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.17 to 0.17], Standard Error of Mean 0.086

26. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Blood Serum: Primary Parameters of Interest (FAS) (IL-8 (pg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 68 | 66
pg/mL | -4.48 (0.929) | -3.92 (0.945)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.6701, ANCOVA; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-3.15 to 2.03], Standard Error of Mean 1.309

27. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Blood Serum: Primary Parameters of Interest (FAS) (MMP Type 9 (ng/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 68 | 66
ng/mL | 0.8 (0.78) | -1.0 (0.79)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.1105, ANCOVA; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-0.4 to 3.9], Standard Error of Mean 1.10

28. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Blood Serum: Primary Parameters of Interest (FAS) (MCP-1(pg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 68 | 66
pg/mL | -24.8 (11.0) | -23.4 (11.21)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.9261, ANCOVA; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-32.4 to 29.5], Standard Error of Mean 15.62

29. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Blood Serum: Primary Parameters of Interest (FAS) (TIMP-1(ng/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 68 | 66
ng/mL | 2.7 (3.19) | -7.5 (3.25)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.0257, ANCOVA; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [1.2 to 19.0], Standard Error of Mean 4.49

30. Secondary Outcome: Change From Baseline of Concentration of Inflammatory Biomarkers in Blood Serum: Primary Parameters of Interest (FAS) (VEGF(pg/mL))
Time Frame: Baseline to 14 weeks
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 68 | 66
pg/mL | 11.3 (12.80) | -21.5 (13.08)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.0728, ANCOVA; Mean Difference (Final Values) = 32.8, 95% CI 2-sided [-3.0 to 168.6], Standard Error of Mean 18.11

31. Secondary Outcome: Change From Baseline in Lung Function Variables: Between-Treatment Differences (FAS) (FEV1 (L))
Time Frame: Baseline to 16 weeks
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 77 | 77
L | 0.028 (0.0212) | -0.035 (0.0212)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.0380, ANCOVA; Mean Difference (Final Values) = 0.063, 95% CI 2-sided [0.004 to 0.122], Standard Error of Mean 0.0300

32. Secondary Outcome: Change From Baseline in Lung Function Variables: Between-Treatment Differences (FAS) (FVC (L))
Time Frame: Baseline to 16 weeks
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 77 | 77
L | 0.031 (0.0391) | -0.033 (0.391)
Statistical Analysis 1: Comparison: R500 vs Placebo; 2-sided 5% test; Test type: Superiority or Other; p = 0.2482, ANCOVA; Mean Difference (Final Values) = 0.064, 95% CI 2-sided [-0.045 to 0.173], Standard Error of Mean 0.0552

33. Secondary Outcome: Wicoxon Signed-rank Test for Change From V2 to V6 in Post-bronchodilator FEV1/FVC
Description: Wilcoxon test is a non-parametric test to evaluate differences among treatments in the variable that is being reported here. The data reported in the outcome measure data table are hodges Lehmann estimate of change from baseline in FEV1/FVC ratio.
Time Frame: Baseline to 16 weeks
Measure: Median (95% Confidence Interval); unit: ratio
Arm/Group | R500 | Placebo
Number analyzed (Participants) | 77 | 77
ratio | 0.5 [0 to 1] | -0.5 [-1 to 0.5]
Statistical Analysis 1: Comparison: R500 vs Placebo; 2 sided 5 % test; Test type: Superiority or Other; p = 0.2629, Wilcoxon (Mann-Whitney); Between treatment difference; Median Difference (Final Values) = -1.00, 95% CI 2-sided [-2.00 to 1.00]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | R500 | Placebo
Serious Adverse Events (participants affected / at risk) | 8/79 | 5/79
Other Adverse Events (participants affected / at risk) | 69/79 | 57/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R500 (N=79) | Placebo (N=79)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Spermatocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R500 (N=79) | Placebo (N=79)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Fatigue (General disorders) | 3 (3) | 3 (3)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 13 (14) | 12 (15)
Rhinitis (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 6 (6) | 2 (2)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Haedache (Nervous system disorders) | 4 (4) | 3 (3)
Lethargy (Nervous system disorders) | 3 (4) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 2 (2)
Bronchial polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
COPD (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No